CLINICAL TRIAL: NCT00757380
Title: Membranepeeling With Trypan Blue Versus Membranpeeling With Brillant Blue for Patients With Idiopathic Epiretinal Membranes
Brief Title: Trypan Blue Versus Brillant Blue for Epiretinal Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Principal Investigator, Dr. Christiane I. Falkner-Radler, MD, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FR-4-CI-2008
Record Dates: First submitted 2008-09-21; First posted 2008-09-23 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Idiopathic Epiretinal Membranes
Keywords: epiretinal membranes; vitreoretinal dyes; membranepeeling
MeSH Terms: conditions — Epiretinal Membrane | interventions — Trypan Blue; procion brilliant blue HGR

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Trypan Blue
  Interventions: Procedure: Trypan Blue
- Group 2 (Active Comparator): Brillant Blue
  Interventions: Procedure: Brillant Blue

INTERVENTIONS:
Procedure: Trypan Blue — Membranepeeling with TB
  Arms: Group 1
Procedure: Brillant Blue — Membranepeeling and membrana limitans interna peeling with BB
  Arms: Group 2

SUMMARY:
Membraneppeling alone versus Membranepeeling with Membrane Limitans Interna Pelling using two different Dyes for Epiretinal Membrane Surgery.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic eperetinal membranes
* Phakic or pseudophakic eyes
* Age over 60 years

Exclusion Criteria:

* Secondary epiretinal membranes
* Severe ocular pathologies

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 3 months

SECONDARY OUTCOMES:
Microperimetry optical coherence tomographie questionnaire (metamorphopsien) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Kreppler, Univ. Doz. Dr., Study Chair — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery; Christiane I Falkner-Radler, Dr., Principal Investigator — The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Locations (1):
- The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery, Vienna, Vienna, Austria